CLINICAL TRIAL: NCT04399655
Title: Highlighting the Medico-economic Interest of an Adapted Physical Activity for Haemodialysis Patients
Acronym: NEPHRACTIVE
Status: Completed | Type: Observational
Sponsor: Clinique Néphrologique Saint-Exupéry (Other)
Responsible Party: Sponsor
Other Study IDs: 01/2020; 2020-A00209-30 (Other: ID-RCB)
Record Dates: First submitted 2020-05-11; First posted 2020-05-22 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-06

CONDITIONS: Chronic Renal Failure; Renal Insufficiency, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic hemodialysis is often associated with a reduction in the quality of life of patients and a reduction in physical activity, due to the repeated frequency of sessions.

Various studies conducted in hemodialysis patients have shown the beneficial effects of physical exercise during hemodialysis sessions on reducing cardiovascular risk, the number of hospitalizations and improving quality of life. It also contributes to improved patient adherence to care.

Finally, it has been shown that exercise during the hemodialysis session is safe for the patient and does not disrupt dialysis parameters.

Nevertheless, there are no data on the medico-economic impact of such a program.

Based on the investigators' experience, the investigators have developed a specific protocol linking the different types of physical activity that have provided evidence of their efficiency and used in standard practice in the investigators' institutions. From tests and questionnaires assessing the physical abilities of patients have already validated for this population in this pathology.

The objective of this project is to show the medico-economic interest of an adapted physical activity program for hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient dependent on the CPAM Haute Garonne,
* Patient affiliated to or beneficiary of a French social security scheme,
* Haemodialysis patient for more than 12 months and in front of benefiting/benefiting from a physical activity program,
* Patient age ≥ at 18 years old,
* French speaking patient.

Exclusion Criteria:

* Patient with cancer, hepatitis, stage 4 arterial disease, arteritis or amputation of a limb
* Pregnant or breastfeeding women according to article L.1121-5 of the CSP,
* Vulnerable persons according to article L.1121-6 of the CSP,
* Persons of full age under guardianship or curatorship or under safeguard of justice,
* Patient unable to personally give his or her consent, or age of majority protected by law,
* Opposition expressed to inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Haemodialysis patient, of full age, for more than 12 months and in front of benefiting/benefiting from a physical activity program
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-04 (Actual)

PRIMARY OUTCOMES:
Variation in direct and indirect medical costs | through study completion, an average of 1 year
  Evaluation of medical costs between the 12 months prior to the start of the adapted physical activity program and the 12 months following the start of the adapted physical activity program.

SECONDARY OUTCOMES:
change in the quality of life score | baseline, at 6 months and at one year
  Assessed by a The Short Form (36) (SF-36 scale) interpreted by an algorythm
change in body mass index, weight and height will be combined to report BMI in kg/m^2 | every month, up to 12 months
  obtained in start of hemodialysis session
change in blood presure in mmHg | every month, up to 12 months
  obtained in start of hemodialysis session
change in rate of haemoglobin in g/dL | every month, up to 12 months
  obtained in start of hemodialysis session
change in percentage of hematocrit and saturation coefficient in % | every month, up to 12 months
  obtained in start of hemodialysis session
change in rate of ferritin in ug/L | every month, up to 12 months
  obtained in start of hemodialysis session
change in rate of urea, transferrin and blood sugar in g/L | every month, up to 12 months
  obtained in start of hemodialysis session
change in rate of potassium in mEq/L | every month, up to 12 months
  obtained in start of hemodialysis session
change in rate of bicarbonate in mmol/L | every month, up to 12 months
  obtained in start of hemodialysis session
change in rate of calcium, phosphore and C-reactiv protein in mg/L | every month, up to 12 months
  obtained in start of hemodialysis session
change in physical activity evaluation score, from 0 (better) to 20 (worse) | baseline, at 6 months and at one year
  obtained thanks to Borg scale

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Néphrologique Saint Saint-Exupéry, Toulouse, France